CLINICAL TRIAL: NCT04276740
Title: Mitochondrial Anti-oxidant Therapy to Resolve Inflammation in Ulcerative Colitis (MARVEL): A Randomised Placebo-controlled Trial on Oral MitoQ in Moderate UC
Brief Title: MARVEL: Mitochondrial Anti-oxidant Therapy to Resolve Inflammation in Ulcerative Colitis
Acronym: MARVEL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: JP Moulton Charitable Foundation (Other); MitoQ (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC19100
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis Flare
MeSH Terms: interventions — mitoquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MitoQ (Active Comparator): Participants will take oral MitoQ 40 mg daily
  Interventions: Dietary Supplement: MitoQ
- Placebo (Placebo Comparator): Participants will take an oral matched placebo daily
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: MitoQ — MitoQ in inflammation: In the experimental setting, MitoQ has been extensively studied with clear mode of action on inflammatory mechanisms relevant to IBD:
  * MitoQ can limit the damage to mitochondria caused by mitochondrial ROS and thereby reducing the leak and oxidisation of mtDNA that are critical to its pro-inflammatory actions within the cell.
  * MitoQ reduces the inflammatory potential of mitochondrial DNA which have escaped or released from dying inflammatory cells.
  * MitoQ can influence how the immune cells generate their energy, diverting it away from a more inflammatory type of metabolism (glycolysis)
  * MitoQ can induce autophagy, a cellular recycling mechanism that removes damaged mitochondria. Defective autophagy is heavily implicated in the pathogenesis of IBD.
  * Hence collectively, MitoQ acts upstream of several pro-inflammatory mechanisms with the net effect to promote resolution of inflammation and mucosal healing.
  Arms: MitoQ
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2b, multi-centered, randomized, placebo-controlled trial with treatment phase over 24 weeks.

Ulcerative Colitis (UC) is a condition that causes inflammation and ulceration of the inner lining of the rectum and colon (the large bowel). In UC, ulcers develop on the surface of the lining and these may bleed and produce mucus. Individuals with UC can become very unwell with disabling bloody diarrhoea, uncontrollable bowel habit and profound tiredness. In very severe cases, UC carry the risks of rupture of the inflamed bowel wall requiring an emergency operation to remove the colon.

The MARVEL study investigates whether MitoQ is a beneficial drug treatment for UC.

Earlier studies have shown that the inflamed UC gut lining releases 'danger signals' arising from the mitochondria. These 'danger signals' attract immune cells and make inflammation worse.

Mitochondria are the 'batteries' or 'power stations' that reside within, and provide energy for living cells. In the gut lining of individuals with UC, the mitochondria are more prone to damage that increases the release of these danger signals.

MitoQ protects the mitochondria and exerts an anti-inflammatory effect. The investigators hypothesise that MitoQ will improve UC and allow the bowels to heal properly following a disease flare.

In the MARVEL study, individuals with an active flare of UC requiring standard oral Prednisolone will be given either MitoQ or placebo as a daily capsule for 24 weeks.

The Investigators will carry out an assessment after 12 and 24 weeks to find out if MitoQ will result in higher rates of improvement in the participants' symptoms and gut lining inflammation. Furthermore, the investigators will investigate if their UC will be better controlled and that they are less likely to need further steroids or more potent forms of drugs.

MitoQ has been shown to be safe in 2 large human clinical studies in Parkinson's disease and Hepatitis C, but the MARVEL study will be the first study in UC. At low doses, MitoQ is used as a nutritional supplement that has an anti-oxidant effect.

Currently, many drug treatments in UC are very strong, expensive and aimed at suppressing the immune system. If the MARVEL study provides supportive data, MitoQ can be a safe and cost-effective new treatment that works at blocking the specific inflammatory signal found in the gut lining of individuals with UC.

ELIGIBILITY:
Inclusion Criteria: • Active UC (Mayo of score 6 or greater with endoscopy subscore of 2 or more); or Partial Mayo Score 4-9 (e.g. without the endoscopic score)

* Baseline rectal bleeding Mayo score of 1 or more
* ≥18 years old
* Confirmed diagnosis of UC confirmed on histology and endoscopic evidence for ≥3 months prior to screening.
* Able to start taking prednisolone at the same time as the study drug/placebo
* Subjects currently receiving the following treatment for UC are eligible providing they have been on stable dose for designated period of time

  * Oral 5-ASA or sulfasalazine stable dose for at least 4 weeks prior to inclusion and during the study period.
  * Azathioprine, 6-mercaptopurine stable dose for 8 weeks prior to study.
  * Topical treatment (5-ASA or steroid based) for active UC flare including suppository and enema.
* Able and willing to give informed consent.

Exclusion Criteria:

* Severe extensive colitis as evidenced by:

  * Physician judgement that the subject is likely to require hospitalisation for medical care or surgical intervention of any kind for UC (e.g. colectomy) within 12 weeks of baseline.
  * Evidence of fulminant colitis, toxic megacolon or recent history of toxic megacolon within the last 6 months; or bowel perforation.
  * Evidence of acute severe UC fulfilling Truelove and Witts Criteria (>6 bloody stools/day with evidence of any of these features: tachycardia [>90bpm], fever [>37.8C], anaemia [Hb <10.5g/dl], low albumin [<30g/l]).
* Any current or previous biologic treatment including anti-TNF therapy or anti-α4β7 therapy; and oral JAK-inhibitors
* Previous treatment for UC, except those listed in the inclusion criteria.
* UC confined to proctitis (distal 15 cm or less)
* UC with Primary Sclerosing Cholangitis (PSC)
* Diagnosis of Crohn's disease or indeterminate colitis
* Pregnancy (Current or attempting to become pregnant during trial period) or breastfeeding
* Cyclosporine, mycophenolate, or tacrolimus administration within 8 weeks of screening.
* Intravenous corticosteroids for treatment of colitis within 8 weeks of screening
* Subjects with current - or recent history of - severe, progressive, or uncontrolled renal, hepatic, haematological, gastrointestinal, metabolic (including uncontrolled hypercholesterolemia), endocrine, pulmonary, cardiac, neurological disease.
* Subjects who have positive stool examinations for enteric pathogens or Clostridium difficile toxin at screening.
* Subjects with a known allergy/contraindication to MitoQ.
* Subjects currently taking any products containing Mitoquinol mesylate (Coenzyme Q10) or any products containing Coenzyme derivatives such as Coenzyme A (CoA, SCoA, CoASH). If subjects are on these products, they can enter the trial after a 7-day washout period.
* Subjects with current barriers in language or communication that in the judgement of local PI will impede the completion of the trial.
* A history of overdose or suicide, or significant active mental health problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2025-12-14 (Actual); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
The proportions of subjects achieving clinical response at Week12 | 12 weeks
  Defined by a decrease from baseline of Mayo Score of at least 3 points and at least 30%, with accompanying decrease in the subscore for rectal bleeding of at least 1 point or an absolute subscore of rectal bleeding of 0 or 1.
  treatment in ulcerative colitis (UC).

SECONDARY OUTCOMES:
Clinical remission at week 12 | 12 weeks
  A complete Mayo score of ≤2 points and no individual subscore >1 point.
Clinical response and remission based on Partial Mayo Score at Week 24 | 24 weeks
  Defined by a Mayo Clinic score of 2 or less + no subscore >1
Longitudinal Analysis of Mucosal healing | 12 weeks
  • Longitudinal Analysis of Mucosal healing - Endoscopic Mayo Score of 0 or 1 at Week 12 and in comparison with baseline Week 0.
Normalization of faecal calprotectin | 24 weeks
  Normalization of faecal calprotectin (<250ug/ml) at week 12 and 24 compared to baseline.
Normalization of faecal haemoglobin | 24 weeks
  Normalization of faecal haemoglobin (<10 ugHb/ g faeces) at week 12 and 24 compared to baseline.
Proportions of participants with primary treatment failure with 24 week study period requiring change in medical treatment as below: | 24 weeks
  * Re-treatment with oral or intravenous corticosteroids
  * Inability to wean off steroids, requiring further increase of Prednisolone during weaning stage due to flare symptoms
  * Biologics (anti-TNF, anti-α4β7, anti-IL23 or Jak-inhibitors)
  * Azathioprine or 6-mercaptopurine in participants who are currently not on a thiopurines
  * Oral or intravenous ciclosporin

CONTACTS AND LOCATIONS:
Overall Officials: David Wilson, MD, Principal Investigator — NHS Lothian
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No